CLINICAL TRIAL: NCT04610424
Title: Cooperative Parent Mediated Therapy in Children With Fragile X Syndrome and Williams Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bambino Gesù Hospital and Research Institute (Other)
Collaborators: Autour Des Williams (Unknown); Acea (Unknown)
Responsible Party: Principal Investigator, Paolo Alfieri, MD, PhD, Bambino Gesù Hospital and Research Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1324_OPBG_2017
Record Dates: First submitted 2020-10-08; First posted 2020-10-30 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Fragile X Syndrome; Williams Syndrome
MeSH Terms: conditions — Fragile X Syndrome; Williams Syndrome

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cooperative Parent Mediated Therapy (Experimental): Cooperative Parent Mediated Therapy" (CPMT) is a targeted parent-mediated intervention focused on the ASD core symptoms (Bearss et al., 2015). CPMT is based on the most significant models of parent training for ASD, in the perspective of Naturalistic Developmental Behavioral Interventions-NDBI with specific attention to the promotion of cooperative interactions (Schreibman et al., 2016). The aim of CPMT is to improve parental skills, to enable parents promoting the following seven target skills in their child: socio-emotional engagement, emotional regulation, imitation, communication, joint attention, play and cognitive flexibility and cooperative interaction. An individualized treatment plan is designed for each child in order to determine his developmental level and treatment goals (Valeri et al., 2019).
  Interventions: Behavioral: Cooperative Parent Mediated Therapy" (CPMT); Behavioral: As usual
- Control (Active Comparator): Control group
  Interventions: Behavioral: As usual

INTERVENTIONS:
Behavioral: Cooperative Parent Mediated Therapy" (CPMT) — CMPT usually last 6 months, for a total amount of 15 sessions of 90 min; twelve core sessions (one session per week) are delivered in the first 3 months, followed by 3 monthly booster sessions. Each weekly core session had a specific focus and specific intervention strategies based on active parent coaching during parent-child interaction, and included the parent-child dyad with the parent being actively coached by a trained therapist. Live active coaching increases parents' competence in implementing strategies to enhance child development, and at the same time increases their confidence. This intervention has demonstrated evidence of effectiveness in socio-communicational improvement as measured by ADOS-G (Valeri, 2019) in a randomized controlled trial (RCT).
  Arms: Cooperative Parent Mediated Therapy
Behavioral: As usual — Speech Language Therapy and Occuapational Therapy provided as usual by National Health Services

SUMMARY:
Fragile X Syndrome (FXS) and Williams-Beuren Syndrome (WBS) are relatively rare disorders characterized by developmental delay associated to socio-communicative deficit and autistic-like behaviours.

WBS has been considered for a long time as the "polar opposite" of ASD, given their hypersociable phenotype. Nonetheless, recent researches have emphasized similarities between ASD and WBS phenotypes. By following some authors "social abnormalities in ASD and WS can be characterized in terms of analogous difficulties in social cognition), and distinct patterns of social motivation which appears to be reduced in ASD and enhanced in WBS". More than opposite condition, these authors suggests that WBS and ASD could share the same difficult in comprehension of social relationship, with opposite pattern of social engagement (enhanced in WBS and weakened ASD). Given, these similarities authors suggest testing the feasibility and validity of therapy for ASD in children with WBS. Parent Mediated Therapy (PMT) is a group of "technique-focused interventions where the parent is the agent of change and the child is the direct beneficiary of treatment". PMT demonstrated evidence of effectiveness in socio-communicational improvement for children with ASD in a randomized controlled trial (RCT).

Some recent researchers have extended the use of PMT to children with genetic disorders and autistic features, such as FXS. While showing encouraging results, the samples of research were limited.

They main aim of this research is to to verify effectiveness of Cooperative PMT (CMPT) for socio-communicative deficit in children with FXS and WBS. Our hypothesis is that CPMT, in addition to conventional rehabilitation therapies (mainly speech therapy and occupational therapies), could contribute to the enhancement of socio-communicative skills and the reduction of behavioural problems. We also expected also an improvement in family quality of life and a reduction of parental stress.

DETAILED DESCRIPTION:
Fragile X Syndrome (FXS) and Williams-Beuren Syndrome (WBS) are relatively rare disorders characterized by developmental delay associated to socio-communicative deficit and autistic-like behaviours. FXS is one of the most common monogenetic cause of syndromic Autism Spectrum Disorder (ASD); up to 60% of males with FXS meet criteria for ASD. Furthermore, around 30%- 35% of children with WBS meet criteria for ASD. WBS has been considered for a long time as the "polar opposite" of ASD, given their hypersociable phenotype and their abnormal interest in social engagement. Nonetheless, recent researches have emphasized similarities between ASD and WBS phenotypes. By following Vivanti "social abnormalities in ASD and WS can be characterized in terms of analogous difficulties in social cognition (the ability to read others' behaviour), and distinct patterns of social motivation (the propensity for social approach/engagement) which appears to be reduced in ASD and enhanced in WS". More than opposite condition, VIvanti suggests that WBS and ASD could share the same difficult in comprehension of social relationship, with opposite pattern of social engagement (enhanced in WBS and weakened ASD). Moreover, some researches showed that children with WS were similarly delayed in global adaptive functioning when compared to ones with ASD. Given, these similarities authors suggest to test the feasibility and validity of therapy for ASD in children with WBS. Parent Mediated Therapy (PMT) is a group of "technique-focused interventions where the parent is the agent of change and the child is the direct beneficiary of treatment". Italian Guidelines for ASD highlight the importance of PMT for ASD treatment. PMT is also strongly recommended by NICE Clinical Guideline CG170 and WHO Mental Health Gap Action Program. PMT has showed evidence of effectiveness in short and long-term symptom reduction in young children with ASD. A research project on the effectiveness of PMT for children with ASD has been activated since 10 years at the Bambino Gesù Children Hospital (BGCH) in Rome. In last years, a semi-manualized intervention called "Cooperative Parent Mediated Therapy" (CPMT) has been systematized. Following Bearss' Parent Training taxonomy, CPMT is a targeted parent-mediated intervention focused on the ASD core symptoms. CPMT is based on the most significant models of parent training for ASD, in the perspective of Naturalistic Developmental Behavioral Interventions-NDBI with specific attention to the promotion of cooperative interactions. The aim of CPMT is to improve parental skills, to enable parents promoting the following seven target skills in their child: socio-emotional engagement, emotional regulation, imitation, communication, joint attention, play and cognitive flexibility and cooperative interaction. An individualized treatment plan is designed for each child in order to determine his developmental level and treatment goals. CMPT usually last 6 months, for a total amount of 15 sessions of 90 min; twelve core sessions (one session per week) are delivered in the first 3 months, followed by 3 monthly booster sessions. Each weekly core session had a specific focus and specific intervention strategies based on active parent coaching during parent-child interaction, and included the parent-child dyad with the parent being actively coached by a trained therapist. Live active coaching increases parents' competence in implementing strategies to enhance child development, and at the same time increases their confidence. This intervention has demonstrated evidence of effectiveness in socio-communicational improvement as measured by ADOS-G in a randomized controlled trial (RCT). On this purpose, some recent researchers have extended the use of PMT to children with genetic disorders and autistic features, such as Fragile X Syndrome (Vismara et al., 2019). While showing encouraging results, the samples of research were limited (four participants); moreover, parent coaching took place mainly through digital services (e.g. video call). Authors suggest implementing RCTs with larger samples in order to evaluate validity of PMT for individuals with FXS. Moreover, as far as we know, there are currently no researches of PMT in patients with WBS.

Since 2017, an experimental, non-pharmacological, randomized, controlled monocentric and non-profit study was started at BGCH in order to verify effectiveness of CPMT for socio-communicative deficit in children with FXS and WBS. Our hypothesis is that CPMT, in addition to conventional rehabilitation therapies (mainly speech therapy and occupational therapies), could contribute to the enhancement of socio-communicative skills and the reduction of behavioural problems. We also expected also an improvement in family quality of life and a reduction of parental stress. The intervention is provided by psychologists with specific training and expertise in CPMT and monitored through supervision by a senior child psychiatrist

Assessment: Children and their family will be evaluated at two time-points, pre randomization (T0) and six months later, at the end of control/treatment period (T1), by means of following assessment tools :

Children: 1. Cognitive Level: Leiter 3/Griffiths III; appropriate tool will be used by evaluation of developmental level 2. Adaptive Level: Vineland Adaptive Behavior Scales, Second Edition; 3. Socio-communication skills: Early Social Communication Scales; the questionnaire Skills Socio-Conversational of the Child (Le abilità socio-conversazionali del bambino; ASCB) ; 4. Language level: Italian adaptation of "MacArthur-Bates Communicative Development Inventories". - Il Primo Vocabolario del Bambino; 5. Behavioural problem: Child Behavior Checklist; 6. Clinical improvement: Clinical Global Impression - Severity scale; Clinical Global Impression - Improvement scale

Parents: 1. Parental Stress: Parenting Stress Index-Short Form; 2. Parental Quality of Life: WHO Quality of Life

ELIGIBILITY:
Inclusion Criteria:

* Molecularly confirmed diagnosis of Fragile X Syndrome
* Molecularly confirmed diagnosis of Williams-Beuren Syndrome
* Autism features
* Score > or = 4 in Clinical Global Impression (Guy et al., 1976)

Exclusion Criteria:

* Parent yet enrolled in a parent training during first evaluation

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Estimated)
Dates: Start 2017-05-17 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Joint attention | 6 months
  Joint attention score from ESCS assessment. Score expressed in percentage of behavior/number of occasion (from 0% to 100%). Higher scores indicate better functioning
Assertivity | 6 months
  Assertivity as measured by Skills Socio-Conversational of the Child. Scores from 1 to 5 (Higher scores indicate better functioning)
Responsivity | 6 months
  Assertivity as measured by Skills Socio-Conversational of the Child. Scores from 1 to 5 (Higher scores indicate better functioning)
Expressive language (Word) | 6 months
  Expressive language as measured by word production scale of Primo vocabolario del bambino (from 0 to 408). higher raw scores indicate higher level of language
Expressive language (Gestures) | 6 months
  Expressive language as measured by gestures production scale of Primo vocabolario del bambino (from 0 to 63). higher raw scores indicate higher level of language
Receptive Language (Word) | 6 months
  Receptive language as measured word comprehension scale of Primo vocabolario del bambino (from 0 to 408). higher raw scores indicate higher level of language
Receptive Language (Sentences) | 6 months
  Receptive language as measured by sentence comprehension scale of Primo vocabolario del bambino (from 0 to 28). higher raw scores indicate higher level of language

SECONDARY OUTCOMES:
Behavioral and emotional problem | 6 months
  Behavioral and emotional problems as measurd by Child Behavior Checklist (T-scores, Mean 50, standard deviation 15). Higher scores indicate severe problems. >64 borderline >70 clinical
Change in Adaptive Level (Vineland Adaptive Behavior Scales, Second Edition) | 6 months
  Adaptive functioning of children. Scores are expressed in standard scores (mean 100, Standard deviation 15). Higher scores indicate better functioning.
Clinical improvement: Clinical Global Impression - Severity scale | 6 months
  Clinical Global Impression - Severity scale is a 7-point scale used to measure baseline severity of patients (Higher scores indicate more severe patient.
Clinical Global Impression - Improvement scale (CGI-I) | 6 months
  Clinical Global Impression - Improvement scale (CGI-I) s a 7-point scale used to measure improvement after treatment (Higher scores indicate more severe symptoms)
Cognitive/developmental Level | 6 months
  Developmental/cognitive level of children as measured by Leiter 3 /Griffiths III. Scores are expressed in standard scores (mean 100, Standard deviation 15). Higher scores indicate better functioning
Quality of Life (Social Relationship) of parents | 6 momths
  Quality of life (Social Relationship) as measured by (WHOQOL). Scores are expressed in raw scores from 0 to 100 (higher scores indicate better quality of life.
Quality of Life (Environmental) of parents | 6 momths
  Quality of life (Environmental) as measured by (WHOQOL). Scores are expressed in raw scores from 0 to 100 (higher scores indicate better quality of life.
Quality of Life (Fisical) of parents | 6 momths
  Quality of life (Fisical) as measured by (WHOQOL). Scores are expressed in raw scores from 0 to 100 (higher scores indicate better quality of life.
Quality of Life (Psychological) of parents | 6 momths
  Quality of life (Psychological) as measured by (WHOQOL). Scores are expressed in raw scores from 0 to 100 (higher scores indicate better quality of life.
Change in Parenting Stress (Parental Distress) | 6 months
  Parenting Stress as measured by Parendal Distress Scale of Parenting Stress Index Short Form. Scores are expressed in percentile (from 5° to 100°). Higher scores indicate higher level of stress
Change in Parenting Stress (Difficult Child) | 6 months
  Parenting Stress as measured by Difficult Child Scale of Parenting Stress Index Short Form. Scores are expressed in percentile (from 5° to 100°). Higher scores indicate higher level of stress
Change in Parenting Stress (Parent-Child Dysfunctional Interaction) | 6 months
  Parenting Stress as measured by Parent-Child Dysfunctional Interaction Scale of Parenting Stress Index Short Form. Scores are expressed in percentile (from 5° to 100°). Higher scores indicate higher level of stress
Change in Parenting Stress (Total Score) | 6 months
  Parenting Stress as measured by Total Stress Scale of Parenting Stress Index Short Form. Scores are expressed in percentile (from 5° to 100°). Higher scores indicate higher level of stress

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Alfieri, PhD, MD, Principal Investigator — Ospedale Pediatrico Bambino Gesù
Locations (1):
- Ospedale Pediatrico Bambino Gesù, Roma, Italy

IPD SHARING:
Plan to Share IPD: No